CLINICAL TRIAL: NCT02660138
Title: A Phase III, Multicentre, Randomised, Double Blind, Parallel Group, Placebo Controlled Study To Assess The Efficacy And Safety Of One Or More Intradetrusor Treatments Of 600 Or 800 Units of Dysport® For The Treatment Of Urinary Incontinence In Subjects With Neurogenic Detrusor Overactivity Due To Spinal Cord Injury Or Multiple Sclerosis
Brief Title: Dysport® Treatment of Urinary Incontinence in Adults Subjects With Neurogenic Detrusor Overactivity (NDO) Due to Spinal Cord Injury or Multiple Sclerosis - Study 1
Acronym: CONTENT1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment of patients
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-FR-52120-222; 2015-003471-30 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 600 U Dysport® Group (Experimental)
  Interventions: Biological: Botulinum toxin type A
- 600 U Dysport® Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo
- 800 U Dysport® Group (Experimental)
  Interventions: Biological: Botulinum toxin type A
- 800 U Dysport® Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 600 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Other Names: AbobotulinumtoxinA (Dysport®); Clostridium BTX-A-haemagglutinin complex
  Arms: 600 U Dysport® Group
Biological: Botulinum toxin type A — 800 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Other Names: AbobotulinumtoxinA (Dysport®); Clostridium BTX-A-haemagglutinin complex
  Arms: 800 U Dysport® Group
Drug: Placebo — AbobotulinumtoxinA Placebo 600 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Arms: 600 U Dysport® Placebo Group
Drug: Placebo — AbobotulinumtoxinA Placebo 800 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Arms: 800 U Dysport® Placebo Group

SUMMARY:
The purpose of this study is to provide confirmatory evidence of the safety and efficacy of two Dysport® (AbobotulinumtoxinA) doses (600 units [U] and 800 U), compared to placebo in reducing urinary incontinence (UI) in adult subjects treated for neurogenic detrusor overactivity (NDO) due to spinal cord injury (SCI) or multiple sclerosis (MS).

ELIGIBILITY:
Key Inclusion Criteria:

* Urinary Incontinence for at least 3 months prior to Screening as a result of Neurogenic Detrusor Overactivity due to Spinal Cord Injury or Multiple Sclerosis.
* Subjects with Spinal Cord Injury must have a stable neurological injury at T1 level or below which occurred at least 6 months prior to Screening.
* Subjects with Multiple Sclerosis must be clinically stable in the investigator's opinion, with no exacerbation (relapse) of MS for at least 3 months prior to Screening.
* Subjects must have had an inadequate response after at least 4 weeks of oral medications used in the treatment of NDO (e.g. anticholinergics, beta-3 agonists) and/or have intolerable side-effects.
* Routinely performing Clean Intermittent Catheterization (CIC) to ensure adequate bladder emptying.
* An average of at least two episodes per day of Urinary Incontinence recorded on the screening bladder diary.

Key Exclusion Criteria:

* Any current condition (other than NDO) that may impact on bladder function.
* Previous or current, tumour or malignancy affecting the spinal column or spinal cord, or any other unstable cause of SCI.
* Any condition that will prevent cystoscopic treatment administration or CIC usage, e.g. urethral strictures.
* Current indwelling bladder catheter, or removal of indwelling bladder catheter less than 4 weeks prior to Screening.
* BTX-A treatment within 9 months prior to Screening for any urological condition (e.g. detrusor or urethral sphincter treatments).
* Any neuromodulation/electrostimulation usage for urinary symptoms/incontinence within 4 weeks prior to Screening. Any implanted neuromodulation device must be switched off at least 4 weeks prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11-09 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (81):
- United States (32):
  - UAB School of Medicine Spain Rehabilitation Center (SRC), Birmingham, Alabama
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Atlantic Urology Medical Group, Long Beach, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Gousse Urology - The Bladder Heath and Reconstructive Urology Institute, Miramar, Florida
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Chesapeake Urology Associates, PA, Owings Mills, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Weill Cornell Medical College, Denville, New Jersey
  - Delaware Valley Urology,IIC, Voorhees Township, New Jersey
  - Urology Group of New Mexico, PC, Albuquerque, New Mexico
  - New York University Langone Medical Center and School of Medicine, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Advanced Urology Centers of New York, Plainview, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Louis Stokes Cleveland Veterans Affairs Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lancaster Urology, Lancaster, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Lahey Hospital & Medical Center, Burlington, Vermont
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Integrity Medical Research, Mountlake Terrace, Washington
  - Medical College of Wisconsin - Freodert Hospital, Milwaukee, Wisconsin
- Canada (4):
  - CHUS - Hôpital Fleurimont, Sherbrooke
  - Sunnybrook Health Sciences Centre, Toronto
  - UBC Hospital - Koerner Pavilion, Vancouver
  - Spinal Cord Research Centre, University of Manitoba, Winnipeg
- Czechia (9):
  - Fakultní Nemocnice Brno, Brno
  - Karlovarska krajska nemocnice, a.s., Karlovy Vary
  - Krajská Nemocnice Liberec, a.s., Liberec
  - Uromedical Center s.r.o., Olomouc
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Thomayerova nemocnice, Prague
  - Fakultní Nemocnice v Motole, Prague
  - Urologicka Ordinace s.r.o., Sternberk
- Italy (6):
  - Azienda Ospedaliero-Universitaria Careggi - Dipartimento Di Neuro-Urologia, Florence
  - Farmacia Istituto Ospedaliero ICOT "Marco Pasquali", Latina
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Perugia
  - Viale Oxford, 81, Roma
  - Ospedale "Bolognini" di Seriate, Seriate
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Udine
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
- Poland (5):
  - Wojewódzki Szpital Zespolony w Elblągu, Elblag
  - Nzoz Neuro-Medic Poradnia Wielospecjalistyczna, Katowice
  - NZOZ Heureka, Piaseczno
  - Szpital Kliniczny Dzieciątka Jezus w Warszawie, Warsaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnią we Wrocławiu, Wroclaw
- Portugal (5):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Alto Ave, EPE, Guimarães
  - British Hospital, Lisbon
  - Centro Hospitalar do Porto, EPE - Hospital Geral de Santo António, Porto
  - Centro Hospitalar de São João, EPE - Hospital de São João, Porto
- Romania (5):
  - Gnosis Evomed, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Fundeni Bucureşti, Bucharest
  - Hifu Terramed Conformal S.R.L, Bucharest
  - Spitalul Clinic Judeţean Mureş, Târgu Mureş
- South Korea (3):
  - 88 Olympic-ro 43-gil, Songpa-gu, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital (UUH), Ulsan
- Turkey (Türkiye) (9):
  - Ankara Üniversitesi Tıp Fakültesi, Ankara
  - Medipol Mega University Hospital, Bağcılar
  - Uludag Universitesi Tip Fakultesi, Uroloji Anabilim Dali, Gorukle, Bursa
  - Marmara Üniversitesi Eğitim ve Araştırma Hastanesi, Istanbul
  - Istanbul Medeniyet Universitesi Goztepe Egitim ve Arastirma Hastanesi Merdivenköy Mah, Istanbul
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri
  - Kocaeli Üniversitesi Tıp Fakültesi, Kocaeli
  - Celal Bayar Universitesi Hafsa Sultan Hastanesi, Manisa
  - Ondokuz Mayıs Üniversitesi Tıp Fakültesi, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Kennelly M, Cruz F, Herschorn S, Abrams P, Onem K, Solomonov VK, Del Rosario Figueroa Coz E, Manu-Marin A, Giannantoni A, Thompson C, Vilain C, Volteau M, Denys P; Dysport CONTENT Program Group. Efficacy and Safety of AbobotulinumtoxinA in Patients with Neurogenic Detrusor Overactivity Incontinence Performing Regular Clean Intermittent Catheterization: Pooled Results from Two Phase 3 Randomized Studies (CONTENT1 and CONTENT2). Eur Urol. 2022 Aug;82(2):223-232. doi: 10.1016/j.eururo.2022.03.010. Epub 2022 Apr 7. PMID 35400537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 227 subjects with urinary incontinence (UI) caused by neurogenic detrusor overactivity (NDO) due to spinal cord injury (SCI) or multiple sclerosis (MS) were randomised at 64 study sites worldwide. One randomised subject was not eligible for entry and did not receive treatment. Hence, 226 subjects were randomised and treated during the study. The study was terminated early by the sponsor due to lack of recruitment.
Pre-assignment Details: Subjects were randomised to 1 of 4 sequences: A) placebo in a double blind placebo controlled (DBPC) cycle then Dysport® 600 Units (U) in subsequent double blind cycles: B) placebo in DBPC cycle then Dysport® 800 U in subsequent cycles: C) Dysport® 600 U in all cycles: D) Dysport® 800 U in all cycles. The minimum re-treatment interval was 12 weeks.
Groups:
- Placebo: Subjects were administered placebo on Day 1 of the DBPC cycle.
  All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 millilitres (mL) divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 600 U: Subjects were administered Dysport® 600 U on Day 1 of the DBPC cycle.
  All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 800 U: Subjects were administered Dysport® 800 U on Day 1 of the DBPC cycle.
  All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
Period: Overall Study
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Started (Subjects randomised in DBPC cycle) | 76 | 76 | 75
Subjects Treated in DBPC Cycle | 76 | 75 | 75
Subjects Entered in the Dysport Cycles | 49 | 75 | 75
Completed (Subjects completed the study in the Dysport cycles) | 6 | 2 | 3
Not Completed | 70 | 74 | 72
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Lack of Efficacy | 1 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 6
Not completed — Lost to Follow-up | 4 | 4 | 1
Not completed — Sponsor Decision to Terminate Study | 57 | 57 | 62
Not completed — Other | 1 | 1 | 0
Not completed — Not treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention to treat (mITT) population: All randomised subjects who received at least 1 administration of study treatment. Subjects were analysed as randomised (planned treatment).
Groups:
- Placebo: Subjects were administered placebo on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 600 U: Subjects were administered Dysport® 600 U for the first study treatment administration on Day 1 of the DBPC cycle.
  All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 800 U: Subjects were administered Dysport® 800 U for the first study treatment administration on Day 1 of the DBPC cycle.
  All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U | Total
Number analyzed (Participants) | 76 | 75 | 75 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 71 | 66 | 205
  >=65 years | 8 | 4 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.15) | 43.0 (12.38) | 46.8 (13.58) | 45.3 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 30 | 95
  Male | 38 | 48 | 45 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 4 | 11
  White | 65 | 70 | 64 | 199
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 3 | 5
Aetiology of NDO [Count of Participants; unit: Participants]
  SCI | 51 | 49 | 48 | 148
  MS | 25 | 26 | 27 | 78

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Weekly Number of UI Episodes at Week 6 of DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The least square (LS) mean of the change in weekly number of UI episodes at 6 weeks after the first study treatment was calculated using a mixed model repeated measures (MMRM) analysis.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: mITT population: All randomised subjects who received at least 1 administration of study treatment. Subjects were analysed as randomised (planned treatment). Only subjects with data available for analysis at Week 6 of DBPC cycle are presented.
Measure: Least Squares Mean (Standard Error); unit: Weekly UI episodes
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 64 | 62 | 67
Weekly UI episodes | -12.7 (2.01) | -23.5 (2.04) | -24.9 (1.97)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, visit (Week 2, Week 6 and Week 12), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [Botulinum toxin [BTX]-naïve or BTX-non-naïve]) and study baseline value (weekly number of UI episodes) as fixed effect variables, and subject as a random effect; Test type: Superiority — If both p-values for the 2 primary tests (the test of Dysport® 800 U vs. placebo and the test of Dysport® 600 U vs. placebo) were lower than 0.05, both were declared statistically significant. If 1 of the primary tests had a p-value greater than or equal to 0.05, then the other test was declared statistically significant if its p-value was lower than 0.025; p = 0.0001, MMRM; LS Mean Difference = -10.83, 95% CI 2-sided [-16.36 to -5.31]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; Treatment group, visit (Week 2, Week 6 and Week 12), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and study baseline value (weekly number of UI episodes) as fixed effect variables, and subject as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, MMRM; LS Mean Difference = -12.19, 95% CI 2-sided [-17.65 to -6.73]

2. Secondary Outcome: Mean Change From Baseline in Maximum Cystometric Capacity (MCC) at Week 6 of DBPC Cycle
Description: All subjects had a standardised urodynamic (filling cystometry) assessment at baseline (screening) and again at Week 6 to determine the MCC. The LS mean of the change in MCC at 6 weeks after the first study treatment was calculated using an analysis of covariance (ANCOVA).
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 66 | 60 | 70
mL | -8.5 (18.06) | 152.4 (19.10) | 180.7 (17.70)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and baseline value of MCC as covariates; Test type: Superiority — This secondary endpoint was included in the hierarchical analysis and was tested for both doses at the 0.05 level using a hierarchical methodology; p < 0.0001, ANCOVA; LS Mean Difference = 160.9, 95% CI 2-sided [109.9 to 211.9]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 189.2, 95% CI 2-sided [140.1 to 238.2]

3. Secondary Outcome: Mean Change From Baseline in Maximum Detrusor Pressure (MDP) at Week 6 of DBPC Cycle
Description: All subjects had a standardised urodynamic filling cystometry assessment at baseline (screening) and again at Week 6 to determine the MDP. The LS mean of the change in MDP at 6 weeks after the first study treatment was calculated using an ANCOVA.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimetres of water
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 58 | 54 | 65
centimetres of water | -5.4 (2.83) | -29.8 (2.96) | -34.1 (2.71)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and baseline value of MDP as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = -24.3, 95% CI 2-sided [-32.3 to -16.4]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = -28.6, 95% CI 2-sided [-36.2 to -21.1]

4. Secondary Outcome: Mean Change From Baseline in Volume at First Involuntary Detrusor Contraction (Vol@1stIDC) at Week 6 of DBPC Cycle
Description: All subjects had a standardised urodynamic (filling cystometry) assessment at baseline (screening) and again at Week 6 to determine the Vol@1stIDC which is the instilled volume when first IDC commences. Subjects who did not exhibit a post-treatment IDC at Week 6 had Vol@1stIDC imputed using the recorded corrected MCC volume at Week 6. The LS mean of the change in Vol@1stIDC at 6 weeks after the first study treatment was calculated using an ANCOVA.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 63 | 56 | 66
mL | 14.0 (19.45) | 169.4 (20.72) | 195.7 (19.12)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and baseline value of Vol@1stIDC as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 155.5, 95% CI 2-sided [100.5 to 210.4]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 181.8, 95% CI 2-sided [129.2 to 234.3]

5. Secondary Outcome: Number of Subjects With No Episodes of UI at Week 6 of DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The number of subjects with no UI episodes at 6 weeks after the first study treatment was recorded and the percentage of subjects was also calculated from the total number of subjects with any number of UI events at Week 6.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: mITT population: All randomised subjects who received at least 1 administration of study treatment . Subjects were analysed as randomised (planned treatment). Only subjects with data available for analysis at Week 6 of DBPC cycle are presented.
Measure: Count of Participants; unit: Participants
Groups:
- Dysport® 800 U: Subjects were administered Dysport® 800 U for on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each.
  Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 64 | 62 | 67
Participants | 3 | 21 | 21
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors, visit (Week 2, Week 6 and Week 12), treatment-by-visit interaction, study baseline-by-visit interaction and study baseline weekly number of UI episodes as fixed effect; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0006, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 9.83, 95% CI 2-sided [2.72 to 35.60]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0003, GLMM; Odds Ratio (OR) = 10.99, 95% CI 2-sided [3.05 to 39.61]

6. Secondary Outcome: Number of Subjects With No IDCs During Storage at Week 6 of DBPC Cycle
Description: All subjects had a standardised urodynamic filling cystometry assessment at baseline (screening) and again at Week 6 to determine the occurrence of IDCs. The number of subjects without IDCs at 6 weeks after the first study treatment was recorded and the percentage of subjects was also calculated from the total number of subjects with data available for analysis at Week 6.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 63 | 60 | 71
Participants | 6 | 20 | 42
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, and recorded stratification factors (aetiology of NDO, previous BTX-A usage) and study baseline (prior intradetrusor BTX-A usage for UI) as explanatory variables; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 5.73, 95% CI 2-sided [2.02 to 16.24]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 6, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 16.08, 95% CI 2-sided [5.82 to 44.43]

7. Secondary Outcome: Mean Change From Baseline in Incontinence Quality of Life (I-QoL) Questionnaire Total Summary Score at Week 6 of DBPC Cycle
Description: The I-QoL questionnaire is a validated, disease-specific questionnaire designed to measure the effect of UI on subjects' QoL. It consists of 22 items in 3 domains (avoidance and limiting behaviour, psychosocial impact and social embarrassment). Subjects used a 5-point response scale for each of the 22 items with values ranging from 1 (extremely) to 5 (not at all). The total summary score was transformed to a 100 point scale ranging from 0 to 100, with higher scores indicating a better QoL. The LS mean of the change in the I-QoL total summary score at 6 weeks after the first study treatment was calculated using a MMRM analysis.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 71 | 61 | 68
score on a scale | 5.8 (2.52) | 19.1 (2.63) | 23.0 (2.51)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, visit (Week 6 and Week 12), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and study baseline value (I-QoL summary total score) as fixed variables, and subject as a random effect; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0003, MMRM; LS Mean Difference = 13.30, 95% CI 2-sided [6.22 to 20.37]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — The secondary endpoint was included in the hierarchical analysis and was tested for both doses at the 0.05 level using a hierarchical methodology; p < 0.0001, MMRM; LS Mean Difference = 17.25, 95% CI 2-sided [10.36 to 24.15]

8. Secondary Outcome: Number of Subjects With a UI Response at Improvement Levels ≥30%, ≥50%, and ≥75% at Week 6 of the DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The number of baseline UI episodes was compared with the number of UI episodes at Week 6 to determine the level of response each subject reached, i.e. a decrease of ≥30%, ≥50% or ≥75% . The number of subjects showing an improvement of ≥30%, ≥50% and ≥75% were recorded and the percentage of subjects was also calculated from the total number of subjects with any number of UI events at Week 6.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 64 | 62 | 67
Participants
  ≥30% Improvement | 32 | 50 | 52
  ≥50% Improvement | 19 | 47 | 50
  ≥75% Improvement | 9 | 39 | 44
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥30% Improvement Level: Dysport® 600 U versus Placebo; Test type: Superiority — Treatment group, recorded stratification factors, visit (Week 2, Week 6 and Week 12), treatment-by-visit interaction, study baseline-by-visit interaction and study baseline weekly number of UI episodes as fixed effect; p = 0.0007, GLMM — This secondary endpoint was not included within the hierarchical testing procedure and was analysed for exploratory purposes only to compare each Dysport® dose to placebo at a 0.05 type one error rate; Odds Ratio (OR) = 4.00, 95% CI 2-sided [1.80 to 8.86]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥30% Improvement Level: Dysport® 800 U versus Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0012, GLMM — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 3.63, 95% CI 2-sided [1.68 to 7.86]
Statistical Analysis 3: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥50% Improvement Level: Dysport® 600 U versus Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 8.03, 95% CI 2-sided [3.56 to 18.09]
Statistical Analysis 4: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥50% Improvement Level: Dysport® 800 U versus Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 8.22, 95% CI 2-sided [3.66 to 18.47]
Statistical Analysis 5: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥75% Improvement Level: Dysport® 600 U versus Placebo; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 10.70, 95% CI 2-sided [4.59 to 24.95]
Statistical Analysis 6: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥75% Improvement Level: Dysport® 800 U versus Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 12.63, 95% CI 2-sided [5.40 to 29.56]

9. Secondary Outcome: Mean Change From Baseline in Volume Per Void at Week 6 of DBPC Cycle
Description: The volume per void was measured during one 24-hour period of the 7-day bladder diary. The LS mean of the change in volume per void at 6 weeks after the first study treatment was calculated using a MMRM analysis.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 62 | 60 | 65
mL | 2.3 (14.92) | 87.1 (15.10) | 112.8 (14.50)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, visit (Week 2, Week 6 and Week 12), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and study baseline value (total volume per void) as fixed effect variables, and subject as a random effect; Test type: Superiority — This secondary endpoint was not included within the hierarchical testing procedure and was analysed for exploratory purposes only to compare each Dysport® dose to placebo at a 0.05 type one error rate; p < 0.0001, MMRM; LS Mean Difference = 84.81, 95% CI 2-sided [43.73 to 125.89]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 9, analysis 1]; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.0001, MMRM; LS Mean Difference = 110.57, 95% CI 2-sided [70.17 to 150.98]

10. Secondary Outcome: Median Time Between Treatments
Description: Duration of effect for time between treatments was calculated by: (the date of the first retreatment visit - date of first treatment administration in the DBPC cycle). The median number of days between treatments was determined based on the Kaplan-Meier method. Subjects with no retreatment were censored at the last visit.
Time Frame: Day of first treatment (baseline) and day of retreatment, up to 2 years
Population: mITT population: All randomised subjects who received at least 1 administration of study treatment. Subjects were analysed as randomised (planned treatment).
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 76 | 75 | 75
days | 120.5 [44 to 616] | 215.0 [37 to 590] | 224.0 [82 to 647]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are presented for the full DBPC cycle (i.e. approximately 35 weeks for both Dysport® groups and approximately 25 weeks for the Placebo group). All cause mortality is presented for the duration of the study (up to a maximum of 113 weeks).
Description: The safety population included all subjects who received at least 1 administration of study treatment (including only partial administration). Safety subjects were analysed according to their actual treatment received. Two subjects randomised to the Dysport 600 U group in the DBPC cycle received Dysport 800 U and are therefore included in the Dysport 800 U group for the safety population.
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/73 | 0/77
Serious Adverse Events (participants affected / at risk) | 8/76 | 9/73 | 6/77
Other Adverse Events (participants affected / at risk) | 23/76 | 20/73 | 23/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Dysport® 600 U (N=73) | Dysport® 800 U (N=77)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (5) | 1 (1)
Appendicitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Dysport® 600 U (N=73) | Dysport® 800 U (N=77)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 13 (26) | 13 (26) | 21 (27)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor on 01 October 2018, due to low subject recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT02660138/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02660138/SAP_001.pdf